CLINICAL TRIAL: NCT02722369
Title: A Phase II, Multicentre, Randomised Trial Comparing Combination Gemcitabine/Carboplatin and Hydroxychloroquine Versus Carboplatin/Etoposide Therapy Alone in Small Cell Lung Cancer (SCLC)
Brief Title: STUDY 15 - Comparing Gemcitabine/Carboplatin and Hydroxychloroquine Versus Carboplatin/Etoposide Therapy Alone in Small Cell Lung Cancer (SCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment, lack of efficacy and increased adverse events in investigational arm.
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCL/12/0515
Record Dates: First submitted 2016-03-08; First posted 2016-03-30 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Gemcitabine; Carboplatin; Etoposide; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): * IV carboplatin AUC5 (area under curve) on Day1
  * IV etoposide 120mg/m2 Day 1, followed by oral etoposide 100mg BD (twice daily) on Day 2 and Day 3
  Interventions: Drug: Carboplatin; Drug: Etoposide
- Investigational Arm (Experimental): * IV gemcitabine 1200mg/m2 on Day 1 and Day 8
  * IV carboplatin AUC5 on Day 1
  * Oral HCQ will be taken at a dose of 400mg BD from day 1 of cycle 1 (maximum of 30 months)
  Interventions: Drug: Gemcitabine; Drug: Carboplatin; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Gemcitabine — Chemotherapy
  Arms: Investigational Arm
Drug: Carboplatin — Chemotherapy
Drug: Etoposide — Chemotherapy
  Arms: Control Arm
Drug: Hydroxychloroquine — Maintenance Agent
  Arms: Investigational Arm

SUMMARY:
To determine whether the combination of gemcitabine/carboplatin with hydroxychloroquine (HCQ) is associated with an improved clinical outcome (progression free and overall survival) compared with chemotherapy alone in patients with small cell lung cancer (SCLC)

DETAILED DESCRIPTION:
This is a multicentre, randomised, phase II trial which aims to compare the combination of hydroxychloroquine and gemcitabine/carboplatin versus standard carboplatin/etoposide chemotherapy, as first line treat in patients with stage IV disease.

The standard first line chemotherapy treatment remains a platinum-based chemotherapy and this has been unchanged for 20 years. Novel active treatment approaches are urgently needed to improve survival in SCLC.

Patients are randomised to one of two treatment arms; carboplatin/etoposide or gemcitabine/carboplatin/hydroxychloroquine.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed SCLC
* Stage IV disease
* Performance status ECOG 0-2
* Life expectancy >8 weeks
* Age 18 or over
* Willing and able to give informed consent
* Patient considered able to tolerate chemotherapy
* Adequate renal function - defined by GFR ≥50mL/min as measured by EDTA or C&G
* Adequate bone marrow reserve: Absolute neutrophil count ≥1.5 x 109/L, haemoglobin ≥90 g/L, platelet count ≥100 x 109/L
* Negative pregnancy test for WCBP
* Highly effective contraception is mandatory for all patients of reproductive potential
* At least one site of measurable disease (target lesion) for RECIST 1.1 evaluation
* Hypersensitivity or history of severe allergic reaction to any of the IMPs
* Able to swallow medication

Exclusion Criteria:

* Mixed cell histology (i.e. NSCLC and SCLC)
* Prior macular degeneration or diabetic retinopathy
* History of glaucoma
* Patients with abnormal LFTs (ALP, ALT/AST*) that are ≥3 x ULN (≥5 x ULN for patients with liver metastases)
* Patients with abnormal bilirubin levels that are ≥1.5 x ULN
* Prior treatment for this disease e.g. chemotherapy, surgery, radiotherapy (except palliative radiotherapy to bone metastases)
* Documented side effects to chloroquine or related agents
* Treatment with chloroquine or related agents within the last year prior to randomisation
* Evidence of significant medical condition or laboratory finding which, in the opinion of the investigator, makes it undesirable for the patient to participate in the trial
* Previous medical history of prolonged QT interval
* A history of prior malignant tumour, unless the patient has been without evidence of disease for at least 3 years or the tumour was a non-melanoma skin tumour or early cervical cancer
* Patients with symptomatic brain metastases
* Women who are breastfeeding
* Concurrent cytochrome P450 enzyme-inducing anticonvulsant drugs e.g. phenytoin, carbamazepine, phenobarbital, primidone or oxcarbazepine
* Patients who are unable to have their digoxin levels regularly monitored

  * if both ALT and AST performed then both need to be recorded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival | Defined as the time from randomisation to first progression/death (whichever came first), assessed up to 41 months

SECONDARY OUTCOMES:
Overall survival | From date of randomisation to death due to any cause, assessed up to 41 months
Objective response as measured by Response Evaluation Criteria in Solid Tumours (RECIST) v.1.1 | From first tumour assessment to progression/trial end (whichever is first), assessed up to 41 months
  Complete Response (CR)/ Partial Response (PR)/ Progressive Disease (PD)/ Stable Disease (SD)
Adverse events | From date of consent to 30 days after final trial treatment
  Including ophthalmologic and treatment specific toxicities
Quality of life as measured by EQ-5D | From baseline to progression/trial end (whichever is first), assessed up to 41 months
  The questionnaire is a standardised questionnaire
Quality of life as measured by QLQC-30 | From baseline to progression/trial end (whichever is first), assessed up to 41 months
  The questionnaire is a standardised questionnaire
Quality of life as measured by QLQ-LC-13 | From baseline to progression/trial end (whicenver is first), assessed up to 41 months
  The questionnaire is a standardised questionnaire
Compliance measured by dose intensity | From first date of trial treatment to progression/trial end (whichever is first), assessed up to 41 months
  Capturing dose delays, modifications and omissions
Compliance measured by dose exposure | From first date of trial treatment to progression/trial end (whichever is first), assessed up to 41 months
  Capturing dose delays, modifications and omissions

CONTACTS AND LOCATIONS:
Locations (13):
- United Kingdom (13):
  - Dorset County Hospital NHS Foundation Trust, Dorchester
  - Royal Surrey County Hospital, Guildford
  - The Princess Alexandra Hospital NHS Trust, Harlow
  - University Hospitals of Morecambe Bay NHS Foundation Trust, Lancaster
  - University Hospital Leicester NHS Trust, Leicester
  - Guy's and St Thomas' Hospitals NHS Foundation Trust, London
  - UCLH, London
  - The Christie, Manchester
  - East and North Herts NHS Foundation Trust, Northwood
  - Nottingham University Hospitals NHS Trust, Nottingham
  - North West Anglia NHS Trust, Peterborough
  - Betsi Cadwaladr University Health Board, Rhyl
  - Airedale NHS Foundation Trust, Steeton

IPD SHARING:
Plan to Share IPD: Yes
On receipt of a request the recipient will consider the proposal, ensure relevant Chief Investigator/Trial Management Group are consulted and, if necessary, Trial Steering Committee and/or Cancer Trials Centre (CTC) Senior Management Group. Any shared data will be in an anonymised format